CLINICAL TRIAL: NCT00973895
Title: VRC 308: An Open-Label Phase I Study of the Safety and Immunogenicity of an Investigational H1 DNA Influenza Vaccine, VRC-FLUDNA057-00-VP, in Healthy Adults 18-70 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 090204; 09-I-0204
Record Dates: First submitted 2009-09-05; First posted 2009-09-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-09-03

CONDITIONS: Influenza A Virus, H1N1 Subtype; Novel Swine-Origin
Keywords: Influenza; Healthy; Immunity; Preventive; Pandemic
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: VRC-FLUDNA057-00-VP — DNA Vaccine Expressing H1 HA from Influenza A/California/04/2009 H1N1 Virus

SUMMARY:
Background:

* Vaccines are substances used to try to create resistance (or immunity) to a disease and to prevent an infection. Researchers are testing a new DNA vaccine designed for a new type of influenza, often referred to as swine flu. The DNA vaccine will instruct the body to make a particular kind of influenza protein that the immune system will be able to recognize.
* Researchers are interested in determining if the vaccine is safe and effective in humans, and would like to study the immune system's response to the vaccine. The vaccine will not give participants influenza; however, it may not be effective in preventing them from getting influenza at a later date.

Objectives:

* To evaluate the safety and tolerability of the VRC-FLUDNA057-00-VP influenza vaccine as administered to healthy adults.
* To evaluate antibody responses to the new influenza vaccine.

Eligibility:

- Healthy adults between the ages of 18 and 70.

Design:

* Participants will have seven planned clinic visits during this study (enrollment day and study weeks 1, 4, 8, 9, 12, and 32).
* All participants will receive three injections of the test vaccine, given as individual doses on day 0, day 28, and day 56 of the study. The vaccine will be given in the upper arm muscle.
* Injections will be given using a needleless system that delivers the vaccine through the skin by using the pressure of carbon dioxide to inject the vaccine through the skin and into the muscle. Participants will remain at the National Institutes of Health (NIH) Clinical Center for at least 30 minutes after the injection to be monitored for any reaction.
* Participants will be asked to keep a 7-day diary card after each injection to record their physical reactions to the vaccine.
* Participants will be asked to return to the NIH Clinical Center as requested by researchers for additional blood tests and other procedures, as required by the study.

DETAILED DESCRIPTION:
STUDY DESIGN- This is an open-label Phase I study to evaluate the safety, tolerability, and immunogenicity of 3- injection vaccination regimen with an investigational plasmid DNA vaccine that encodes for H1 hemagglutinin (HA) of an H1N1 influenza virus. All study participants will be offered to receive an additional optional booster immunization with licensed inactivated monovalent H1N1 influenza vaccine.

The hypothesis is that the DNA vaccine will be safe for human administration and will elicit an antibody response. The primary objectives are to evaluate the safety and tolerability of the VRC-FLUDNA057-00-VP DNA vaccine at a dosage of 4 mg administered in a 3-injection schedule. The secondary objectives are to evaluate antibody responses including induced antibody titer as measured by a hemagglutination inhibition (HAI) assay and to document the reactogenicity of the inactivated H1N1 influenza vaccine when administered to subjects previously vaccinated with the VRC-FLUDNA057-00-VP DNA vaccine.

Exploratory objectives are related to further evaluation of the humoral and cellular immune responses, including the responses after each injection and after the boost with licensed H1N1 inactivated influenza vaccine.

PRODUCT DESCRIPTIONS- The VRC-FLUDNA057-00-VP vaccine was developed and manufactured by VRC, NIAID and is composed of 1 closed-circular DNA plasmid with a CMV/R promoter that encodes for the H1 hemagglutinin from the Influenza A/California/04/2009 H1N1 virus, identified late in the 2008-2009 northern hemisphere (NH) influenza season that has been referred to as swine flu in news reports. Vaccine vials will be supplied at 4 mg/mL and each 4 mg dosage will require a 1 mL injection. Vaccinations with the H1 DNA vaccine will be administered intramuscularly (IM) in the deltoid muscle using the Biojector[R] 2000 Needle-Free Injection Management System (Biojector). Licensed inactivated monovalent H1N1 influenza vaccine will be obtained through the NIH Clinical Center (CC) pharmacy, for use as a booster injection, and administered with needle and syringe. The brand administered will depend upon what is available through the NIH CC.

SUBJECTS- A total of 20 healthy adults in the 18-70 years age range will be enrolled; however, no more than 10 subjects will be in the 51-70 year old age range.

STUDY PLAN- All subjects will receive 3 injections of the H1 DNA vaccine as shown in the schedule below. No more than 5 subjects may be enrolled in the first week of the study. Following the 5th enrollment, the remainder of subjects may be enrolled without restrictions on enrollment rate. All subjects that have no contraindications to the licensed - inactivated H1N1 influenza vaccine or to additional blood drawing will be offered the option to receive the licensed inactivated H1N1 influenza vaccine. The study includes 7 clinic visits and 3 telephone contacts as well as 3 additional visits for subjects that opt to receive an inactivated influenza vaccine. Subjects who have received the inactivated H1N1 vaccine outside of the VRC Clinic after Study Week 12 may consent to contribute the additional research samples through completing the extra visits on the schedule for post boost evaluations. A target window for the inactivated H1N1 vaccine is shown in the schema below. However, given that all subjects will be at or beyond Study Week 12, the earliest mutually convenient date after the H1N1 vaccine supply and amended protocol become available is acceptable for administration of the optional injection. The added post-boost research sample collections will then be scheduled to occur relative to the date the H1N1 booster injection.

Number of Subjects = 20

VRC-FLUDNA057-00-VP 4 mg on Day 0; 4mg on Day 28 plus or minus 7; 4mg on Day 56 plus or minus 7, at least 21 days between injections. Inactivated licensed H1N1 influenza vaccine (optional) Day 168 plus or minus 28 - 1 dose

STUDY DURATION- Each participant will complete 32 weeks of clinical follow up.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18 to 70 years old.
  2. Available for clinical follow-up through Week 32.
  3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
  4. Complete an AoU prior to enrollment and verbalize understanding of all questions answered incorrectly.
  5. Able and willing to complete the informed consent process.
  6. Willing to donate blood for sample storage to be used for future research.
  7. No evidence of previously undiagnosed clinically significant chronic diseases.
  8. Physical examination and laboratory results without clinically significant findings, no fever (greater than or equal to 100.4 degree F) in the 72 hours prior to enrollment, and a Body Mass Index (BMI) greater than or equal to 18 and < 42 within the 56 days prior to enrollment.

     Laboratory Criteria within 56 days prior to enrollment:
  9. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men
  10. White blood cells (WBC) = 3,300-12,000 cells/mm(3)
  11. Differential either within institutional normal range or accompanied by site physician approval as a differential that is consistent with healthy volunteer status
  12. Total lymphocyte count greater than or equal to 800 cells/mm(3)
  13. Platelets = 125,000 - 500,000/mm(3)
  14. Alanine aminotransferase (ALT) less than or equal to 2.5 times upper limit of normal (ULN)
  15. Serum creatinine less than or equal to 1 times ULN (less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males) and estimated glomerular filtration rate > 60 mL/min/1.73 m(2).
  16. Negative FDA-approved HIV blood test. [Note: Results of HIV enzyme-linked immunosorbent assay (ELISA) will be documented, but a negative HIV polymerase chain reaction (PCR) test result will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study].

      Female-Specific Criteria:
  17. Negative human chorionic gonadotropin (HCG) pregnancy test (urine or serum) for women presumed to be of reproductive potential on the day of enrollment.
  18. A female subject must meet one of the following criteria:

      No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

      OR

      Agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 32 of the study,

      OR

      Agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 32 of the study by one of the following methods:

      (Bullet) condoms, male or female, with or without a spermicide;

      (Bullet) diaphragm or cervical cap with spermicide;

      (Bullet) intrauterine device;

      (Bullet) contraceptive pills, patch, implant or any other FDA-approved contraceptive method;

      (Bullet) male partner has previously undergone a vasectomy.

      EXCLUSION CRITERIA

      Women Specific:

  <!-- -->

  1. Breast-feeding or planning to become pregnant during the first 32 weeks after enrollment in the study.

     Subject has received any of the following substances:
  2. Systemic immunosuppressive medications or cytotoxic medications within the 12 weeks prior to enrollment. [With the exceptions that a short course (duration of 10 days or less or a single injection) of corticosteroids for a self-limited condition at least 2 weeks prior to enrollment in this study will not exclude study participation.]
  3. Blood products within 112 days (16 weeks) prior to HIV screening
  4. Immunoglobulin within 56 days (8 weeks) prior to HIV screening
  5. Live attenuated vaccines within 28 days (4 weeks) prior to initial study vaccine administration
  6. Investigational research agents within 28 days (4 weeks) prior to initial study vaccine administration
  7. Medically indicated subunit or killed vaccines (e.g., pneumococcal, or allergy treatment with antigen injections) within 14 days (2 weeks) of initial study vaccine administration
  8. Current anti-TB prophylaxis or therapy

     Subject has a history of any of the following clinically significant conditions:
  9. Serious reactions to vaccines that preclude receipt of study vaccinations as determined by investigator.
  10. Hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
  11. Asthma that is severe, unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral, intravenous, or high dose inhaled corticosteroids.
  12. Diabetes mellitus type I.
  13. Thyroid disease that is not well-controlled.
  14. Generalized idiopathic urticaria within the last 1 year.
  15. Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.

  16 Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.

  17. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.

  18. Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years.

  19. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.

  20. Guillain-Barr Syndrome.

  21.Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide plan or attempt.

  22. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08-06; Primary Completion 2010-09-03 (Actual); Study Completion 2010-09-03 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity, lab tests, AEs) | 32 weeks

SECONDARY OUTCOMES:
Immunogenicity (cellular and humoral immune function assays) | 32 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Subbarao K, Murphy BR, Fauci AS. Development of effective vaccines against pandemic influenza. Immunity. 2006 Jan;24(1):5-9. doi: 10.1016/j.immuni.2005.12.005. PMID 16413916
- [Background] Luke CJ, Subbarao K. Vaccines for pandemic influenza. Emerg Infect Dis. 2006 Jan;12(1):66-72. doi: 10.3201/eid1201.051147. PMID 16494720
- [Background] Karron RA, Callahan K, Luke C, Thumar B, McAuliffe J, Schappell E, Joseph T, Coelingh K, Jin H, Kemble G, Murphy BR, Subbarao K. A live attenuated H9N2 influenza vaccine is well tolerated and immunogenic in healthy adults. J Infect Dis. 2009 Mar 1;199(5):711-6. doi: 10.1086/596558. PMID 19210163
- [Derived] Crank MC, Gordon IJ, Yamshchikov GV, Sitar S, Hu Z, Enama ME, Holman LA, Bailer RT, Pearce MB, Koup RA, Mascola JR, Nabel GJ, Tumpey TM, Schwartz RM, Graham BS, Ledgerwood JE; VRC 308 Study Team. Phase 1 study of pandemic H1 DNA vaccine in healthy adults. PLoS One. 2015 Apr 17;10(4):e0123969. doi: 10.1371/journal.pone.0123969. eCollection 2015. PMID 25884189